CLINICAL TRIAL: NCT06774001
Title: A Global Prospective Cohort Study on Outcomes of Appendicectomy for Appendicitis
Acronym: AlliGatOr
Status: Recruiting | Type: Observational
Sponsor: University of Birmingham (Other)
Collaborators: Christian Medical College and Hospital, Ludhiana, India (Other); Ministry of Health, Ghana (Other Government); Lagos University Teaching Hospital (LUTH) (Unknown); Hospital Español Veracruz (Unknown); WITS Health Consortium (South Africa) (Unknown); University of Abomey Calavi, Benin (Unknown); Kigali University Teaching Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AL_20241016
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Appendicitis; Appendectomy
Keywords: Appendicectomy; Appendicitis; Appendectomy
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Appendicectomy for suspected or confirmed appendicitis: All patients undergoing appendicectomy for suspected or confirmed appendicitis by any surgical approach should be included. This includes patients who went theatre with suspect appendicitis even if the intraoperative or pathology results found a different diagnosis, so long as an appendicectomy was performed. It also includes patients who went to theatre for reasons other than suspected appendicitis but were found to have appendicitis intraoperatively and underwent appendicectomy. This includes interval appendicectomy and right hemicolectomy if performed for acute appendicitis.
  There are no age restrictions, although, if appropriate participating hospitals can choose to only include children or only adults, based on an age cut-off of their choice.
  Interventions: Procedure: Appendicectomy

INTERVENTIONS:
Procedure: Appendicectomy — Both open and minimally invasive (laparoscopic and robotic) interventions are eligible for inclusion. Laparoscopic and robotic converted to open cases are also eligible.

SUMMARY:
This study aims to assess and improve the global management of appendicitis, the most common emergency surgery, by examining various aspects of emergency care systems worldwide. Appendicitis is a time-sensitive condition, and delays in diagnosis or treatment can lead to complications, affecting patient outcomes and increasing healthcare costs. The study uses appendicitis as a "tracer condition" to explore how different healthcare systems manage emergency care, focusing on factors like access, quality, and efficiency. By gathering data from hospitals worldwide, the study seeks to identify areas where emergency surgical care can be improved, particularly in low- and middle-income countries (LMICs).

The main goal is to identify gaps in emergency care systems, using a set of key performance measures (KPMs) that assess access to care, the quality of surgical treatment, and patient safety. These include factors like the time from symptom onset to first surgical assessment, the rate of appendectomy performed via minimally invasive (laparoscopic) surgery, and postoperative complications. The study aims to collect data on at least 14,000 patients from around 500 hospitals globally between February and May 2025. The data will be analyzed by hospital income group (from low to high) to understand how different resource levels impact outcomes and to help guide future policy and practice improvements.

The study also includes two sub-studies that focus on specific issues in surgical care. The Sustainability and Waste Management sub-study aims to explore how hospitals manage waste and sustainability practices in operating theatres. This sub-study is part of global efforts to reduce carbon emissions in healthcare settings. The Financing sub-study examines the financial burden of appendicectomy, particularly the out-of-pocket costs for patients in LMICs. It will explore how the costs of open vs. laparoscopic surgery differ and investigate the impact of these costs on patients.

By combining global data on clinical outcomes with information on hospital resources and patient finances, this study hopes to provide valuable insights into how to improve emergency surgical care across diverse settings, making recommendations that can lead to better access to safe, timely, and affordable treatment for appendicitis worldwide.

DETAILED DESCRIPTION:
This prospective, multicentre, global cohort study will capture patients within an overall study window of 3 February 2025 to 25 May 2025. Any hospital performing appendicectomy worldwide will be eligible to participate, collecting data over 14 days for consecutive patients undergoing appendicectomy for suspected or confirmed acute appendicitis.

The primary aim is to identify areas for system strengthening in emergency surgery using appendicitis as a tracer condition with a pre-defined key performance measurement set. The secondary aims of this study are to evaluate variations in the presentation, diagnosis, management, access to minimally invasive surgery, and outcomes of patients that have surgery for suspected acute appendicitis. Variation could be assessed across groups stratified by human development index, hospital funding, urban/rural, and facility level.

All consecutive patients undergoing appendicectomy for suspected or confirmed appendicitis are eligible for inclusion and should be captured in the study. No additional follow-up is required for this study. Follow-up data will be collected from routine health records.

Based on previous NIHR-GSU prospective cohort studies, this study is anticipated to include around 500 hospitals. Based on an average of one appendectomy per day and two 14-day data collection blocks per hospital, we anticipate capturing data for 14,000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: There are no age restrictions, although, if appropriate participating hospitals can choose to only include children or only adults, based on an age cut-off of their choice.
* Procedure: All patients undergoing appendicectomy for suspected or confirmed appendicitis by any surgical approach should be included. This includes patients who went theatre with suspect appendicitis even if the intraoperative or pathology results found a different diagnosis, so long as an appendicectomy was performed. It also includes patients who went to theatre for reasons other than suspected appendicitis but were found to have appendicitis intraoperatively and underwent appendicectomy. This includes interval appendicectomy and right hemicolectomy if performed for acute appendicitis.
* Approach: Both open and minimally invasive (laparoscopic and robotic) interventions are eligible for inclusion. Laparoscopic and robotic converted to open cases are also eligible.

Exclusion Criteria:

* Indication: Appendicectomy for any indication other than suspected or confirmed appendicitis should be excluded. For example, patients having appendicectomy for known appendiceal neoplasm.
* Procedure: Patients having appendectomy as part of another surgical procedure should be excluded. For example, patients having removal of appendix as part of a colon cancer procedure are not eligible for inclusion.
* Approach: Natural orifice surgery and endoscopic treatment for suspected appendicitis are excluded.
* Previous appendicectomy: Patients having surgery for stump appendicitis are excluded.
* Return to theatre: Patients should be entered into study only once. A patient returning to theatre after appendectomy should not be re-entered as a new patient.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients undergoing appendicectomy for suspected or confirmed appendicitis are eligible for inclusion and should be captured in the study.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time from symptom onset to first assessment by the surgical team | Any time up to point of first assessment by surgical team
  Duration from onset of symptoms to first assessment by the surgical team
Perforation rate | Within 30 days postoperatively
  Proportion of all patients with histology-confirmed appendicitis who had a perforated appendix on histology
Imaging | From presentation to time of Surgery
  Proportion of all patients having preoperative cross-sectional (CT/MRI) imaging
Laparoscopy rate | Time from Knife to Skin to end of operation
  Proportion of all patients undergoing a laparoscopic approach for appendicectomy
Time from first assessment to theatre | Time from first assessment by surgical team to knife on skin
  Duration from decision to operate to knife to skin
Negative appendicectomy rate | Within 30 days postoperatively
  Proportion of all patients with a histologically normal appendix
Post-operative length of stay | Within 30 days postoperatively
  Length of stay (in days) in hospital after appendicectomy. Day of surgery is considered day 0.
30-day overall Clavien-Dindo complications | Within 30 days postoperatively
  Adverse post-operative events may be classified in different ways:
  * Failure of treatment
  * Sequelae
  * Complication Definitions of these are provided in Appendix C of the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Aneel Bhangu, Study Director — University of Birmingham
Locations (7):
- University of Abomey Calavi, Cotonou, Benin
- Tamale Teaching Hospital, Tamale, Ghana
- Christian Medical College and Hospital Ludhiana, Ludhiana, India
- Hospital Espanol Veracruz, Veraruz, Mexico
- Lagos University Teaching Hospital, Lagos, Nigeria
- University Teaching Hospital of Kigali (CHUK), Kigali, Rwanda
- Chris Hani Baragwanath Academic Hospital, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No
Alligator is collecting only routinely collected hospital data, seeking to measure current clinical practice.